CLINICAL TRIAL: NCT01202760
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of LY2127399 in Patients With Rheumatoid Arthritis (RA) With or Without Background Disease-Modifying Anti-rheumatic Drug (DMARD) Therapy (FLEX O)
Brief Title: A Rheumatoid Arthritis Study in Participants
Acronym: FLEX O
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12978; H9B-MC-BCDO (Other: Eli Lilly and Company); CTRI/2011/07/001867 (Registry Identifier: Clinical Trials Registry India)
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Results first posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tabalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 120 mg LY2127399 (Experimental): LY2127399: 120 milligrams (mg), subcutaneous (SC) injection, every 4 weeks for 24 weeks. Participants received a 240-mg (2 SC injections of 120 mg each) loading dose of LY2127399 when initiating treatment.
  During the Treatment Period, for blinding purposes, participants alternated injections of LY2127399 and injections of Placebo every 2 weeks.
  After 16 weeks, non-responders received 90 mg of LY2127399 every 2 weeks for the rest of the 24-week Treatment Period.
  Interventions: Drug: LY2127399; Drug: Placebo
- 90 mg LY2127399 (Experimental): LY2127399: 90 milligrams (mg), subcutaneous (SC) injection, every 2 weeks for 24 weeks. Participants received a 180-mg (2 SC injections of 90 mg each) loading dose of LY2127399 when initiating treatment.
  After 16 weeks, non-responders continued to receive 90 mg of LY2127399 every 2 weeks for the rest of the 24-week Treatment Period.
  Interventions: Drug: LY2127399
- Placebo (Placebo Comparator): Placebo: subcutaneous (SC) injection, every 2 weeks for 24 weeks. Participants received a loading dose of 2 SC injections of Placebo when initiating treatment.
  After 16 weeks, non-responders received 90 milligrams (mg) of LY2127399 every 2 weeks for the rest of the 24-week Treatment Period.
  Interventions: Drug: LY2127399; Drug: Placebo

INTERVENTIONS:
Drug: LY2127399
  Other Names: Tabalumab
Drug: Placebo
  Arms: 120 mg LY2127399; Placebo

SUMMARY:
The primary purpose of this study is to help answer if LY2127399 is safe and effective in the treatment of rheumatoid arthritis with or without background disease-modifying anti-rheumatic drug (DMARD) therapy.

This study is comprised of 2 periods:

Period 1 - 24-week blinded treatment

Period 2 - 48-week post-treatment follow-up

DETAILED DESCRIPTION:
In consideration of disease severity, all participants were assessed for non-response at Week 16. A total of 66 joints were examined for swelling, and a total of 66 joint were examined for tenderness. For participants who had at least 5 swollen and 5 tender joints at baseline, Week 16 non-responders (NRs) were defined as participants with <20% improvement from baseline in both tender joint counts and swollen joint counts. For participants who did not have at least 5 swollen and 5 tender joints at baseline, Week 16 NRs were defined as participants who had at least 2 additional tender and 2 additional swollen joints from baseline. All Week 16 NRs and all participants who discontinued study treatment at any time, for any reason, were defined as NRs starting at that timepoint and going forward for all American College of Rheumatology (ACR) imputed analyses, including the Week 24 endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis (RA) of more than 6 months and less than 15 years
* Global Assessment of Disease Activity visual analog scale (VAS) greater than or equal to 20/100 millimeters (mm)
* If on one or more conventional disease-modifying anti-rheumatic Drugs (DMARDs) at randomization, must have been on a stable dose for at least 8 weeks prior to study start.
* Women must not be pregnant, breastfeeding, or become pregnant during the study

Exclusion Criteria:

* Use of unstable doses of non-steroidal inflammatory drugs (NSAIDS) in the past 6 weeks
* Steroid injection or intravenous (IV) infusion in the last 6 weeks
* Use of more than 10 milligrams per day (mg/day) of oral steroids in the last 6 weeks
* Use of biologic DMARD concurrently or recently
* History of a serious reaction to other biological DMARDs
* Use of an oral calcineurin inhibitor (for example, cyclosporin or tacrolimus) in the last 8 weeks
* Surgery on a joint or other major surgery less than 2 months prior to study start, or plans to have joint surgery or major surgery during the study
* Active fibromyalgia, juvenile chronic arthritis, spondyloarthropathy, Crohn's disease, ulcerative colitis, psoriatic arthritis, or other systemic inflammatory condition except RA
* Cervical cancer or squamous skin cancer within the past 3 years, or other cancer within the past 5 years
* Received a live vaccine within the past 12 weeks (for example, vaccines for measles, mumps, rubella, and chicken pox, and nasal-spray flu vaccines)
* Hepatitis or human immunodeficiency virus (HIV)
* A serious bacterial infection (for example, pneumonia or cellulitis) within 3 months or a serious bone or joint infection within 6 months
* Symptoms of herpes zoster or herpes simplex within the last month
* Active or latent tuberculosis (TB)
* Current symptoms of a serious disorder or illness
* Use of an investigational drug within the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1004 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (213):
- United States (77):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paradise Valley, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hot Springs, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrance, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Whittier, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wildomar, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colorado Springs, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lewes, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aventura, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeBary, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Harbor, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pinellas Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. Petersburg, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tamarac, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Venice, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zephyrhills, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Decatur, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lawrenceville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Savannah, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eagle, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morton Grove, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockford, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cumberland, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyannis, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Worcester, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bingham Farms, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Clair Shores, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flowood, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jackson, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lincoln, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roslyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Syracuse, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hickory, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bend, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethlehem, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Limerick, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pottstown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Myrtle Beach, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Jackson, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubbock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesquite, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nassau Bay, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Richland Hills, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sugar Land, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
- Argentina (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mar del Plata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kogarah, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herston, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malvern East
- Bulgaria (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burgas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pleven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plovdiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rousse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sevlievo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sofia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Varna
- Colombia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bogotá
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Medellín
- Croatia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Opatija
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rijeka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Split
- Hungary (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiskunhalas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nyíregyháza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sátoraljaújhely
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szikszó
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Veszprém
- India (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahmedabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chennai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaipur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mysore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nellore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Delhi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Secunderabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Surat
- Japan (22):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mie
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ohita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sapporo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tomakomai
- Lithuania (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alytus
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaunas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Klaipedos
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Šiauliai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vilnius
- Malaysia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Batu Caves
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuantan Pahang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perak
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sarawak
- Mexico (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aguascalientes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexicali
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morelia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Querétaro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tijuana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tlalpan
- New Zealand (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotorua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tauranga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timaru
- Poland (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdynia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ploieşti
- Russia (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barnaul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kemerovo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kursk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nizhny Novgorod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Novosibirsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ryazan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stavropol
- Slovakia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Piešťany
- South Africa (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Benoni
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloemfontein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Breyten
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cape Town
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durban
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Limpopo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pretoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Somerset West
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stellenbosch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westville
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Busan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Sri Lanka (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colombo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalubowila
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nugegoda
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Keelong
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuei Shan Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- Ukraine (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dnipropetrovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kharkiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiev
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odesa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poltava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Simferopol
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vinnytsia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Started | 379 | 374 | 251
Received at Least One Dose of Study Drug | 379 | 371 | 250
Completed | 332 | 322 | 216
Not Completed | 47 | 52 | 35
Not completed — Entry Criteria Not Met | 0 | 3 | 1
Not completed — Adverse Event | 11 | 9 | 10
Not completed — Death | 2 | 1 | 0
Not completed — Lack of Efficacy | 6 | 8 | 7
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Parent / Caregiver Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 17 | 18 | 14
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Protocol Violation | 7 | 5 | 2
Not completed — Sponsor Decision | 4 | 4 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants, including participants who did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo | Total
Number analyzed (Participants) | 379 | 374 | 251 | 1004
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (11.2) | 50.6 (12.2) | 51.0 (12.0) | 51.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 293 | 295 | 209 | 797
  Male | 86 | 79 | 42 | 207
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 47 | 24 | 109
  Not Hispanic or Latino | 193 | 185 | 133 | 511
  Unknown or Not Reported | 148 | 142 | 94 | 384
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13 | 21 | 9 | 43
  Asian | 96 | 93 | 59 | 248
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 12 | 13 | 14 | 39
  White | 254 | 235 | 162 | 651
  More than one race | 2 | 9 | 6 | 17
  Unknown or Not Reported | 1 | 2 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 126 | 125 | 83 | 334
  Argentina | 7 | 6 | 5 | 18
  Colombia | 9 | 9 | 5 | 23
  Mexico | 20 | 25 | 15 | 60
  Bulgaria | 13 | 13 | 12 | 38
  Croatia | 2 | 1 | 3 | 6
  Hungary | 3 | 12 | 6 | 21
  Lithuania | 14 | 10 | 11 | 35
  Poland | 27 | 22 | 12 | 61
  Romania | 0 | 1 | 3 | 4
  Russia | 14 | 13 | 8 | 35
  Slovakia | 8 | 3 | 2 | 13
  Ukraine | 16 | 15 | 6 | 37
  Australia | 2 | 3 | 2 | 7
  India | 14 | 9 | 9 | 32
  Japan | 44 | 42 | 28 | 114
  South Korea | 7 | 6 | 5 | 18
  Malaysia | 2 | 4 | 1 | 7
  New Zealand | 6 | 2 | 6 | 14
  Sri Lanka | 4 | 4 | 2 | 10
  South Africa | 32 | 38 | 24 | 94
  Taiwan | 9 | 11 | 3 | 23
Tender Joint Count (68 Count) [Mean (Standard Deviation); unit: joint count] — Tender joint count is the number of tender and painful joints determined for each participant by examination of 68 joints. Joints were assessed by pressure and joint manipulation on physical examination. Participants were asked for pain sensations on these manipulations and watched for spontaneous pain reactions. Any positive response on pressure, movement, or both is translated into a single tender-versus-nontender dichotomy.
  joint count | 22.8 (15.5) | 23.7 (17.1) | 22.8 (15.2) | 23.2 (16.0)
Swollen Joint Count (66 Count) [Mean (Standard Deviation); unit: joint count] — Swollen joint count is the number of swollen joints determined for each participant by examination of 66 joints. Joints were classified as either swollen or not swollen. Swelling was defined as palpable fluctuating synovitis of the joint.
  joint count | 14.8 (11.6) | 15.3 (11.6) | 14.3 (10.6) | 14.8 (11.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology 20% (ACR20) Response
Description: ACR20 Responder Index: Composite of clinical, laboratory, and functional measures of rheumatoid arthritis. ACR20 Responder: had >=20% improvement from baseline in both 68 tender and 66 swollen joint counts and >=20% improvement in at least 3 of 5 criteria: participant's and physician's global assessment of disease activity, Health Assessment Questionnaire-Disability Index (HAQ-DI) (which measured participants' perceived degree of difficulty performing daily activities), joint pain, and C-reactive protein (CRP). Percentage of participants achieving ACR20 response=(number of ACR20 responders/number of participants treated)*100. All non-responders at Week 16 as well as all participants who discontinued study treatment at any time, for any reason, were defined as non-responders starting at that timepoint and going forward, including Week 24 endpoint.
Time Frame: Up to 24 weeks
Population: All randomized participants with at least 5/68 tender joints and 5/66 swollen joints at baseline and with evaluable ACR20 data. If participant's CRP was missing, last postbaseline value was used. If ACR was missing after carrying forward CRP, last postbaseline ACR response was used. Data after Week 16 for Week 16 non-responders was not included.
Measure: Number; unit: percentage of participants
Groups:
- 120 mg LY2127399: LY2127399: 120 milligrams (mg), subcutaneous (SC) injection, every 4 weeks for 24 weeks. Participants received a 240 mg (2 SC injections of 120 mg each) loading dose when initiating treatment.
- 90 mg LY2127399: LY2127399: 90 milligrams (mg), subcutaneous (SC) injection, every 2 weeks for 24 weeks. Participants received a 180 mg (2 SC injections of 90 mg each) loading dose when initiating treatment.
- Placebo: Placebo: subcutaneous (SC) injection, every 2 weeks for 24 weeks. Participants received a loading dose of 2 SC injections when initiating treatment.
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 320 | 316 | 213
percentage of participants | 34.4 | 33.5 | 31.5

2. Secondary Outcome: Percentage of Participants With American College of Rheumatology 50% (ACR50) and 70% (ACR70) Responses
Description: ACR Responder Index: Composite of clinical, laboratory, and functional measures of rheumatoid arthritis. ACR50 Responder: had >=50% improvement from baseline in both 68 tender joint (TJ) and 66 swollen joint (SJ) counts and >=50% improvement in at least 3/5 criteria: participant's (Pt's) and physician's global assessment of disease activity, HAQ-DI (measured Pts' perceived degree of difficulty performing daily activities), joint pain, and CRP. Percentage of Pt achieving ACR50 response=(number (No) of ACR50 responders/No of Pts treated)*100. ACR70 Responder: had >=70% improvement from baseline in both TJ and SJ counts and >=70% improvement in at least 3 of same 5 criteria for ACR50. Percentage of Pts achieving ACR70 response=(No of ACR70 responders/No of Pts treated)*100. All non-responders at Week 16 as well as all Pts who discontinued study treatment at any time, for any reason, were defined as non-responders starting at that timepoint and going forward, including Week 24 endpoint.
Time Frame: Up to 24 weeks
Population: All randomized participants with at least 5/68 TJ and 5/66 SJ at baseline and with evaluable ACR50 or ACR70 responder data. If participant's CRP was missing, last postbaseline value was used. If ACR was missing after carrying forward CRP, last postbaseline ACR response was used. Data after Week 16 for Week 16 non-responders was not included.
Measure: Number; unit: percentage of participants
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 320 | 316 | 213
percentage of participants
  ACR50 | 11.6 | 11.7 | 12.7
  ACR70 | 4.7 | 6.3 | 4.7

3. Secondary Outcome: Mean Percent Improvement in American College of Rheumatology Percent Improvement (ACR-N)
Description: ACR-N is a continuous measure of clinical, laboratory, and functional outcomes in rheumatoid arthritis that characterizes percentage of improvement in disease activity from baseline based on ACR core set. Percentage of improvement was truncated to range of -100 to 100 to minimize impact of outliers (greater values indicate greater percent improvement). This index was calculated as minimum of a) percentage of improvement in TJ count, b) percentage of improvement in SJ count, or c) third highest percentage of improvement of remaining 5 ACR core criteria: If >=3 components of the 5 ACR core criteria were missing, then c) was set to missing; if any of 3 components a), b), or c) were missing, then ACR-N was set to missing. Least Squares (LS) means were calculated using analysis of covariance (ANCOVA) with treatment, region, tumor necrosis factor-inadequate responder treatment history, and disease-modifying anti-rheumatic drug (DMARD) background as fixed factors and baseline as a covariate.
Time Frame: Up to 24 weeks
Population: All randomized participants with at least 5/68 tender joints and at least 5/66 swollen joints at baseline and with evaluable ACR-N data. Modified last observation carried forward (mLOCF) was used to impute missing postbaseline values. Data after Week 16 for Week 16 non-responders was not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 318 | 314 | 211
units on a scale | -11.5 (4.6) | -9.5 (4.6) | -11.5 (5.0)

4. Secondary Outcome: Change From Baseline to 24 Weeks in Tender Joint Count (68 Joint Count)
Description: Tender joint count is the number of tender and painful joints determined for each participant by examination of 68 joints. Joints were assessed by pressure and joint manipulation on physical examination. Participants were asked for pain sensations on these manipulations and watched for spontaneous pain reactions. Any positive response on pressure, movement, or both is translated into a single tender-versus-nontender dichotomy. LS means were calculated using ANCOVA with treatment, region, tumor necrosis factor-inadequate responder treatment history, and DMARD background as fixed factors and baseline as a covariate.
Time Frame: Baseline, up to 24 weeks
Population: All randomized participants with at least 5/68 tender joints and at least 5/66 swollen joints at baseline and with evaluable tender joint count data. Modified last observation carried forward (mLOCF) was used to impute missing postbaseline values. Data after Week 16 for Week 16 non-responders was not included.
Measure: Least Squares Mean (Standard Error); unit: joint count
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 318 | 315 | 211
joint count | -1.61 (1.30) | -1.63 (1.31) | -2.11 (1.40)

5. Secondary Outcome: Change From Baseline to 24 Weeks in Swollen Joint Count (66 Joint Count)
Description: Swollen joint count is the number of swollen joints determined for each participant by examination of 66 joints. Joints were classified as either swollen or not swollen. Swelling was defined as palpable fluctuating synovitis of the joint. LS means were calculated using ANCOVA with treatment, region, tumor necrosis factor-inadequate responder treatment history, and DMARD background as fixed factors and baseline as a covariate.
Time Frame: Baseline, up to 24 weeks
Population: All randomized participants with at least 5/68 tender joints and at least 5/66 swollen joints at baseline and with evaluable swollen joint count data. Modified last observation carried forward (mLOCF) was used to impute missing postbaseline values. Data after Week 16 for Week 16 non-responders was not included.
Measure: Least Squares Mean (Standard Error); unit: joint count
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 318 | 315 | 211
joint count | -2.59 (0.97) | -3.18 (0.99) | -3.59 (1.05)

6. Secondary Outcome: Change From Baseline to 24 Weeks in Participant's Assessment of Pain (Visual Analog Scale)
Description: Participant's assessment of their current arthritis pain using a visual analog scale (VAS) ranged from 0 millimeters (mm) (no pain) to 100 mm (worst possible pain). A decrease in pain score indicated an improvement in the participant's condition. LS means were calculated using ANCOVA with treatment, region, tumor necrosis factor-inadequate responder treatment history, and DMARD background as fixed factors and baseline as a covariate.
Time Frame: Baseline, up to 24 weeks
Population: All randomized participants with at least 5/68 tender joints and at least 5/66 swollen joints at baseline and with evaluable participant's assessment of pain data. Modified last observation carried forward (mLOCF) was used to impute missing postbaseline values. Data after Week 16 for Week 16 non-responders was not included.
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 313 | 312 | 208
millimeters | -9.0 (2.3) | -9.6 (2.4) | -6.9 (2.5)

7. Secondary Outcome: Change From Baseline to 24 Weeks in Participant's Global Assessment of Disease Activity (Visual Analog Scale)
Description: Participant's assessment of their current arthritis disease activity using a visual analog scale (VAS) ranged from 0 millimeters (mm) (no arthritis activity) to 100 mm (extremely active arthritis). A decrease in disease activity score indicated an improvement in the participant's condition. LS means were calculated using ANCOVA with treatment, region, tumor necrosis factor-inadequate responder treatment history, and DMARD background as fixed factors and baseline as a covariate.
Time Frame: Baseline, up to 24 weeks
Population: All randomized participants with at least 5/68 tender joints and at least 5/66 swollen joints at baseline and with evaluable participant's global assessment of disease activity data. Modified last observation carried forward (mLOCF) was used to impute missing postbaseline values. Data after Week 16 for Week 16 non-responders was not included.
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 317 | 313 | 211
millimeters | -10.2 (2.3) | -10.2 (2.4) | -6.9 (2.5)

8. Secondary Outcome: Change From Baseline to 24 Weeks in Physician's Global Assessment of Disease Activity (Visual Analog Scale)
Description: Physician's assessment of the participant's current arthritis disease activity using a visual analog scale (VAS) ranged from 0 millimeters (mm) (no arthritis activity) to 100 mm (extremely active arthritis). A decrease in disease activity score indicated an improvement in the participant's condition. LS means were calculated using ANCOVA with treatment, region, tumor necrosis factor-inadequate responder treatment history, and DMARD background as fixed factors and baseline as a covariate.
Time Frame: Baseline, up to 24 weeks
Population: All randomized participants with at least 5/68 tender joints and at least 5/66 swollen joints at baseline and with evaluable physician's global assessment of disease activity data. Modified last observation carried forward (mLOCF) was used to impute missing postbaseline values. Data after Week 16 for Week 16 non-responders was not included.
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 308 | 306 | 201
millimeters | -10.0 (2.3) | -12.4 (2.4) | -9.7 (2.5)

9. Secondary Outcome: Change From Baseline to 24 Weeks in Disease Activity Score (Based on 28 Joint Count)-C-Reactive Protein (DAS28-CRP)
Description: Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), C-reactive protein (CRP) (milligrams per liter), and participant global assessment of disease activity using visual analog scale (VAS) (participant global VAS). DAS28-CRP was calculated using following formula: DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*participant global VAS+0.96. Scores ranged 1.0-9.4, where lower scores indicated less disease activity and remission is DAS28-CRP <2.6. A decrease in DAS28-CRP indicated an improvement in participant's condition. LS means were calculated using ANCOVA with treatment, region, tumor necrosis factor-inadequate responder treatment history, and DMARD background as fixed factors and baseline as a covariate.
Time Frame: Baseline, up to 24 weeks
Population: All randomized participants, even if participant did not take assigned treatment, did not receive correct treatment, or otherwise did not follow protocol, with evaluable DAS28-CRP data. Modified last observation carried forward (mLOCF) was used to impute missing postbaseline values. Data after Week 16 for Week 16 non-responders was not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 376 | 369 | 249
units on a scale | -0.42 (0.12) | -0.49 (0.12) | -0.41 (0.13)

10. Secondary Outcome: Change From Baseline to 24 Weeks in Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: The HAQ-DI questionnaire assesses the participant's self-perception on the degree of difficulty [0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do)] when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area, which ranged from 0 (no disability) to 3 (severe disability), were averaged to calculate HAQ-DI. A decrease in HAQ-DI score indicated an improvement in the participant's condition. LS means were calculated using ANCOVA with treatment, region, tumor necrosis factor-inadequate responder treatment history, and DMARD background as fixed factors and baseline as a covariate.
Time Frame: Baseline, up to 24 weeks
Population: All randomized participants with at least 5/68 tender joints and at least 5/66 swollen joints at baseline and with evaluable HAQ-DI data. Modified last observation carried forward (mLOCF) was used to impute missing postbaseline values. Data after Week 16 for Week 16 non-responders was not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 317 | 314 | 211
units on a scale | -0.21 (0.05) | -0.18 (0.05) | -0.15 (0.05)

11. Secondary Outcome: Time to American College of Rheumatology 20% (ACR20) Response
Description: ACR20 Responder Index: Composite of clinical, laboratory, and functional measures of rheumatoid arthritis. ACR20 Responder: had >= 20% improvement from baseline in both 68 tender and 66 swollen joint counts and >=20% improvement in at least 3 of 5 criteria: participant's and physician's global assessment of disease activity, Health Assessment Questionnaire-Disability Index (HAQ-DI) (which measured participants' perceived degree of difficulty performing daily activities), joint pain, and C-reactive protein (CRP). The Kaplan-Meier estimator was used to summarize time to ACR20 response over the Treatment Period (24 weeks). The time to American College of Rheumatology 20% (ACR20) response (in weeks) is calculated as:
  (Date of the first postbaseline visit during the Treatment Period meeting ACR20 response criteria - Date of first injection of study treatment + 1) / 7.
Time Frame: Baseline through 24 weeks
Population: All randomized participants with at least 5/68 tender joints and at least 5/66 swollen joints at baseline and with evaluable ACR20 response data. Week 16 non-responders were counted as responders if they responded prior to Week 16. Otherwise, they were censored at the date of the Week 16 injection.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- 120 mg LY2127399: LY2127399: 120 milligrams (mg), subcutaneous (SC) injection, every 4 weeks for 24 weeks. Participants received a 240 mg (2 SC injections of 120 mg each) loading dose when initiating treatment.
  After 16 weeks, non-responders received 90 mg every 2 weeks for the rest of the 24-week Treatment Period.
- 90 mg LY2127399: LY2127399: 90 milligrams (mg), subcutaneous (SC) injection, every 2 weeks for 24 weeks. Participants received a 180 mg (2 SC injections of 90 mg each) loading dose when initiating treatment.
  After 16 weeks, non-responders continued to receive 90 mg every 2 weeks for the rest of the 24-week Treatment Period.
- Placebo: Placebo: subcutaneous (SC) injection, every 2 weeks for 24 weeks. Participants received a loading dose of 2 SC injections when initiating treatment.
  After 16 weeks, non-responders received 90 milligrams (mg) of LY2127399 every 2 weeks for the rest of the 24-week Treatment Period.
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 318 | 315 | 210
weeks | 16.7 [16.1 to 20.1] | 16.1 [12.1 to 20.1] | 16.4 [15.9 to 23.6]

12. Secondary Outcome: Probability of an ACR20 Response by 24 Weeks
Description: as for outcome 11
Time Frame: Baseline through 24 weeks
Population: as for outcome 11
Measure: Number; unit: probability of response
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 318 | 315 | 210
probability of response | 0.612 | 0.611 | 0.608

13. Secondary Outcome: Percentage of Participants With DAS28-Based European League Against Rheumatism (EULAR) Response
Description: EULAR Responder index based on 28 joint count categorizes clinical response based on improvement since baseline in DAS28-CRP. Participants are categorized as EULAR responders or non-responders based on improvement of DAS28-CRP scores from baseline. EULAR28 responder is defined as either DAS28-CRP <=5.1 and DAS28-CRP change <-0.6; or DAS28-CRP >5.1 and DAS28-CRP change <-1.2. EULAR28 responder index is defined as good response: DAS28-CRP <=3.2 and DAS28-CRP change <-1.2; moderate response: DAS28-CRP change <-1.2 except cases defined in good response; or DAS28-CRP <=5.1 and DAS28-CRP change <-0.6 and >-1.2. EULAR Remission is defined as a DAS28-CRP score of <2.6.
Time Frame: Up to 24 weeks
Population: All randomized participants with at least 5/68 tender joints and at least 5/66 swollen joints at baseline and with evaluable EULAR response data. Modified last observation carried forward (mLOCF) was used to impute missing postbaseline values. Data after Week 16 for Week 16 non-responders was not included.
Measure: Number; unit: percentage of participants
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 318 | 314 | 211
percentage of participants | 50.3 | 49.7 | 46.4

14. Secondary Outcome: Change From Baseline to 24 Weeks in Medical Outcomes Study 36-Item Short Form (SF-36) Health Status Survey Domain and Summary Scores
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and 2 component scores (mental [MCS] and physical health [PCS]). Domain scores calculated by summing each item for each domain and transforming scores into 0-100 scale; higher scores indicated better health status. MCS score consisted of social functioning, vitality, mental health, and role-emotional scales. PCS score consisted of physical functioning, bodily pain, role-physical, and general health scales. LS means were calculated using ANCOVA with treatment, region, tumor necrosis factor-inadequate responder treatment history, and DMARD background as fixed factors and baseline as a covariate.
Time Frame: Baseline, up to 24 weeks
Population: All randomized participants with at least 5/68 tender joints and at least 5/66 swollen joints at baseline and with evaluable SF-36 domain and summary scores. Modified last observation carried forward (mLOCF) was used to impute missing postbaseline values. Data after Week 16 for Week 16 non-responders was not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 311 | 304 | 206
units on a scale
  Physical functioning domain | 2.07 (0.84) | 3.14 (0.85) | 1.48 (0.91)
  Bodily pain domain | 1.62 (0.82) | 2.08 (0.83) | 1.34 (0.89)
  Role limitations due to physical problems domain | 1.60 (0.83) | 2.40 (0.84) | 1.65 (0.91)
  Role limitations due to emotional problems domain | 3.30 (1.01) | 3.23 (1.02) | 3.11 (1.09)
  General health perception domain | 1.93 (0.76) | 1.99 (0.77) | 1.81 (0.82)
  Mental health domain | 3.09 (0.89) | 3.00 (0.90) | 2.31 (0.97)
  Social function domain | 1.17 (1.00) | 1.24 (1.01) | 0.33 (1.08)
  Vitality domain | 2.85 (0.87) | 2.58 (0.88) | 2.22 (0.94)
  Physical component summary score | 1.19 (0.79) | 2.10 (0.79) | 1.14 (0.85)
  Mental component summary score | 3.18 (0.95) | 2.68 (0.96) | 2.54 (1.03)

15. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) up to Week 24 Endpoint
Description: CRP is an indicator of inflammation. A negative change indicated an improvement in the participant's condition. LS means were calculated using ANCOVA with treatment, region, tumor necrosis factor-inadequate responder treatment history, and DMARD background as fixed factors and baseline as a covariate.
Time Frame: Baseline, up to 24 weeks
Population: All randomized participants with at least 5/68 tender joints and 5/66 swollen joints at baseline and with evaluable CRP data. Modified last observation carried forward (mLOCF) was used to impute missing postbaseline values. Data after Week 16 for Week 16 non-responders was not included.
Measure: Least Squares Mean (Standard Error); unit: milligrams per liter (mg/L)
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 318 | 315 | 211
milligrams per liter (mg/L) | 2.69 (1.42) | 1.92 (1.44) | 1.76 (1.54)

16. Secondary Outcome: Change From Baseline to 24 Weeks in Absolute CD3-CD20+ B-cell Counts
Description: Cell-surface marker cluster designation (CD) 3 negative, CD20 positive (CD3-CD20+) defines total mature B cells. B-lymphocyte antigen CD20 is an activated-glycosylated phosphoprotein expressed on the surface of all mature B cells. Baseline B-cell count is determined by calculating the average of the 2 pretreatment B-cell counts obtained once during Days -28 through -7 and on Day 0. A positive or negative change indicated an increase or decrease, respectively in B-cell count. LS means were calculated using ANCOVA with treatment, region, tumor necrosis factor-inadequate responder treatment history, and DMARD background as fixed factors and baseline as a covariate.
Time Frame: Baseline, up to 24 weeks
Population: All randomized participants who received at least 1 dose of study treatment with evaluable absolute B-cell data. Modified last observation carried forward (mLOCF) was used to impute missing postbaseline values. Data after Week 16 for Week 16 non-responders was not included.
Measure: Least Squares Mean (Standard Error); unit: cells per microliter
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 376 | 370 | 248
cells per microliter | -50.5 (19.4) | -74.4 (19.3) | -0.7 (20.9)

17. Secondary Outcome: Change From Baseline to 24 Weeks in Serum Immunoglobulin (Ig) Levels
Description: Immunoglobulins, or antibodies, are large proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. Change from baseline serum immunoglobulin G (IgG), immunoglobulin A (IgA), and immunoglobulin M (IgM) levels are reported. A negative change indicated a decrease in immunoglobulin levels. LS means were calculated using ANCOVA with treatment, region, tumor necrosis factor-inadequate responder treatment history, and DMARD background as fixed factors and baseline as a covariate.
Time Frame: Baseline, up to 24 weeks
Population: All randomized participants who received at least 1 dose of study treatment with evaluable serum immunoglobulin (Ig) data. Modified last observation carried forward (mLOCF) was used to impute missing postbaseline values.
Measure: Least Squares Mean (Standard Error); unit: grams per liter (g/L)
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 374 | 369 | 248
grams per liter (g/L)
  Immunoglobulin G | -0.813 (0.165) | -0.758 (0.165) | 0.117 (0.178)
  Immunoglobulin A | -0.209 (0.044) | -0.224 (0.044) | 0.139 (0.047)
  Immunoglobulin M | -0.267 (0.026) | -0.275 (0.025) | -0.049 (0.028)

18. Secondary Outcome: Population Pharmacokinetics (PK)
Description: Population estimate of constant clearance as determined by population pharmacokinetics (PK) analysis. A 2-compartment model was used in PK modeling.
Time Frame: Baseline through 24 weeks
Population: Participants who received at least 1 dose of LY2127399 with evaluable LY2127399 PK data.
Measure: Mean (95% Confidence Interval); unit: milliliter per hour (mL/h)
Groups:
- LY2127399: 120 milligrams (mg) LY2127399: subcutaneous (SC) injection, every 4 weeks for 24 weeks. Participants received a 240 mg (2 SC injections of 120 mg each) loading dose when initiating treatment.
  90 milligrams (mg) LY2127399: subcutaneous (SC) injection, every 2 weeks for 24 weeks. Participants received a 180 mg (2 SC injections of 90 mg each) loading dose when initiating treatment.
  After 16 weeks, non-responders received 90 mg every 2 weeks for the rest of the 24-week Treatment Period.
Arm/Group | LY2127399
Number analyzed (Participants) | 777
milliliter per hour (mL/h) | 3.60 (2.54) [3.44 to 3.78]

19. Secondary Outcome: Percentage of Participants Developing Anti-LY2127399 Antibodies
Description: LY2127399 anti-drug antibodies (ADA) were assessed at baseline, 1, 4, 16, and 24 weeks. Percentage of participants (Pts) with ADA=(number of Pts with treatment-emergent ADA/number of Pts assessed)*100. Pts with treatment-emergent ADA were Pts who had any sample from baseline up to and through Week 24 that was a 4-fold increase (2-dilution increase) in immunogenicity titer over baseline titer, or Pts who tested negative at baseline and positive post-baseline (at titer of ≥1:20).
Time Frame: Baseline through 24 weeks
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 376 | 370 | 248
percentage of participants | 2.4 | 1.9 | 2.8

ADVERSE EVENTS:
Groups:
- 120 mg LY2127399, Randomized Treatment Period: LY2127399: 120 milligrams (mg), subcutaneous (SC) injection, every 4 weeks for 24 weeks. Participants received a 240 mg (2 SC injections of 120 mg each) loading dose when initiating treatment.
  During the Treatment Period, for blinding purposes, participants alternated injections of LY2127399 and injections of placebo every 2 weeks.
  The Randomized Treatment Period was defined as the time all data was collected during the Treatment Period, excluding the data collected after the date of the Week 16 injection for the Week 16 non-responders.
- 90 mg LY2127399, Randomized Treatment Period: LY2127399: 90 milligrams (mg), subcutaneous (SC) injection, every 2 weeks for 24 weeks. Participants received a 180 mg (2 SC injections of 90 mg each) loading dose when initiating treatment.
  The Randomized Treatment Period was defined as the time all data was collected during the Treatment Period, excluding the data collected after the date of the Week 16 injection for the Week 16 non-responders.
- Placebo, Randomized Treatment Period: Placebo: subcutaneous (SC) injection, every 2 weeks for 24 weeks. Participants received a loading dose of 2 SC injections when initiating treatment.
  The Randomized Treatment Period was defined as the time all data was collected during the Treatment Period, excluding the data collected after the date of the Week 16 injection for the Week 16 non-responders.
- 120 mg LY2127399, Rescue Period: LY2127399: 120 milligrams (mg), subcutaneous (SC) injection, every 4 weeks for 24 weeks. Participants received a 240 mg (2 SC injections of 120 mg each) loading dose when initiating treatment.
  During the Treatment Period, for blinding purposes, participants alternated injections of LY2127399 and injections of placebo every 2 weeks.
  After 16 weeks, non-responders received 90 mg every 2 weeks for the rest of the 24-week Treatment Period.
  The Rescue Treatment Period was defined as all data collected after the date of the Week 16 injection during the Treatment Period for Week 16 non-responders.
- 90 mg LY2127399, Rescue Period: LY2127399: 90 milligrams (mg), subcutaneous (SC) injection, every 2 weeks for 24 weeks. Participants received a 180 mg (2 SC injections of 90 mg each) loading dose when initiating treatment.
  After 16 weeks, non-responders continued to receive 90 mg every 2 weeks for the rest of the 24-week Treatment Period.
  The Rescue Treatment Period was defined as all data collected after the date of the Week 16 injection during the Treatment Period for Week 16 non-responders.
- Placebo, Rescue Period: Placebo: subcutaneous (SC) injection, every 2 weeks for 24 weeks. Participants received a loading dose of 2 SC injections when initiating treatment.
  After 16 weeks, non-responders received 90 milligrams (mg) of LY2127399 every 2 weeks for the rest of the 24-week Treatment Period.
  The Rescue Treatment Period was defined as all data collected after the date of the Week 16 injection during the Treatment Period for Week 16 non-responders.
- 120 mg LY2127399, Follow-up Period: LY2127399: 120 milligrams (mg), subcutaneous (SC) injection, every 4 weeks for 24 weeks. Participants received a 240 mg (2 SC injections of 120 mg each) loading dose when initiating treatment.
  During the Treatment Period, for blinding purposes, participants alternated injections of LY2127399 and injections of placebo every 2 weeks.
  The Post-Treatment Follow-Up Period started after Week 24 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
- 90 mg LY2127399, Follow-up Period: LY2127399: 90 milligrams (mg), subcutaneous (SC) injection, every 2 weeks for 24 weeks. Participants received a 180 mg (2 SC injections of 90 mg each) loading dose when initiating treatment.
  The Post-Treatment Follow-Up Period started after Week 24 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
- Placebo, Follow-up Period: Placebo: subcutaneous (SC) injection, every 2 weeks for 24 weeks. Participants received a loading dose of 2 SC injections when initiating treatment.
  The Post-Treatment Follow-Up Period started after Week 24 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
- 120 mg LY2127399 to 90 mg LY212739 (Week 16), Follow-up Period: LY2127399: 120 milligrams (mg), subcutaneous (SC) injection, every 4 weeks for 24 weeks. Participants received a 240 mg (2 SC injections of 120 mg each) loading dose when initiating treatment.
  During the Treatment Period, for blinding purposes, participants alternated injections of LY2127399 and injections of placebo every 2 weeks.
  After 16 weeks, non-responders received 90 mg every 2 weeks for the rest of the 24-week Treatment Period.
  The Post-Treatment Follow-Up Period started after Week 24 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
- Placebo to 90 mg LY2127399 (Week 16), Follow-up Period: Placebo: subcutaneous (SC) injection, every 2 weeks for 24 weeks. Participants received a loading dose of 2 SC injections when initiating treatment.
  After 16 weeks, non-responders received 90 milligrams (mg) of LY2127399 every 2 weeks for the rest of the 24-week Treatment Period.
  The Post-Treatment Follow-Up Period started after Week 24 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
Arm/Group | 120 mg LY2127399, Randomized Treatment Period | 90 mg LY2127399, Randomized Treatment Period | Placebo, Randomized Treatment Period | 120 mg LY2127399, Rescue Period | 90 mg LY2127399, Rescue Period | Placebo, Rescue Period | 120 mg LY2127399, Follow-up Period | 90 mg LY2127399, Follow-up Period | Placebo, Follow-up Period | 120 mg LY2127399 to 90 mg LY212739 (Week 16), Follow-up Period | Placebo to 90 mg LY2127399 (Week 16), Follow-up Period
Serious Adverse Events (participants affected / at risk) | 14/379 | 8/371 | 7/250 | 5/81 | 0/72 | 0/56 | 0/40 | 4/45 | 3/37 | 1/7 | 2/12
Other Adverse Events (participants affected / at risk) | 174/379 | 154/371 | 98/250 | 23/81 | 16/72 | 9/56 | 12/40 | 17/45 | 13/37 | 5/7 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 120 mg LY2127399, Randomized Treatment Period (N=379) | 90 mg LY2127399, Randomized Treatment Period (N=371) | Placebo, Randomized Treatment Period (N=250) | 120 mg LY2127399, Rescue Period (N=81) | 90 mg LY2127399, Rescue Period (N=72) | Placebo, Rescue Period (N=56) | 120 mg LY2127399, Follow-up Period (N=40) | 90 mg LY2127399, Follow-up Period (N=45) | Placebo, Follow-up Period (N=37) | 120 mg LY2127399 to 90 mg LY212739 (Week 16), Follow-up Period (N=7) | Placebo to 90 mg LY2127399 (Week 16), Follow-up Period (N=12)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/293 (0) | 0/292 (0) | 0/208 (0) | 0/61 (0) | 0/60 (0) | 0/42 (0) | 0/31 (0) | 0/35 (0) | 1/27 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/293 (1) | 0/292 (0) | 0/208 (0) | 0/61 (0) | 0/60 (0) | 0/42 (0) | 0/31 (0) | 0/35 (0) | 0/27 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0/293 (0) | 1/292 (1) | 0/208 (0) | 0/61 (0) | 0/60 (0) | 0/42 (0) | 0/31 (0) | 0/35 (0) | 0/27 (0) | 0 (0) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1/293 (1) | 0/292 (0) | 0/208 (0) | 0/61 (0) | 0/60 (0) | 0/42 (0) | 0/31 (0) | 0/35 (0) | 0/27 (0) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0/293 (0) | 0/292 (0) | 1/208 (1) | 0/61 (0) | 0/60 (0) | 0/42 (0) | 0/31 (0) | 0/35 (0) | 0/27 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 120 mg LY2127399, Randomized Treatment Period (N=379) | 90 mg LY2127399, Randomized Treatment Period (N=371) | Placebo, Randomized Treatment Period (N=250) | 120 mg LY2127399, Rescue Period (N=81) | 90 mg LY2127399, Rescue Period (N=72) | Placebo, Rescue Period (N=56) | 120 mg LY2127399, Follow-up Period (N=40) | 90 mg LY2127399, Follow-up Period (N=45) | Placebo, Follow-up Period (N=37) | 120 mg LY2127399 to 90 mg LY212739 (Week 16), Follow-up Period (N=7) | Placebo to 90 mg LY2127399 (Week 16), Follow-up Period (N=12)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macular pigmentation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 6 (7) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 8 (10) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (9) | 8 (10) | 6 (8) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 5 (5) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 4 (9) | 10 (27) | 2 (3) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 8 (10) | 11 (34) | 2 (2) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 7 (7) | 10 (10) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 14 (14) | 9 (9) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 4 (4) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 17 (20) | 14 (16) | 9 (10) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 5 (5) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 6 (6) | 11 (12) | 6 (6) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 12 (15) | 28 (29) | 10 (12) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (8) | 4 (5) | 6 (8) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/293 (0) | 1/292 (1) | 0/208 (0) | 0/61 (0) | 0/60 (0) | 0/42 (0) | 0/31 (0) | 0/35 (0) | 1/27 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 6 (6) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Computerised tomogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin d decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 6 (6) | 8 (9) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 9 (9) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 17 (17) | 10 (12) | 13 (13) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 12 (12) | 5 (7) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 16 (17) | 13 (16) | 6 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 2 (2) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2/293 (2) | 0/292 (0) | 0/208 (0) | 0/61 (0) | 0/60 (0) | 0/42 (0) | 1/31 (1) | 0/35 (0) | 0/27 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 7 (7) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 10 (10) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balanitis (Reproductive system and breast disorders) | 0/86 (0) | 0/79 (0) | 0/42 (0) | 0/20 (0) | 0/12 (0) | 0/14 (0) | 0/9 (0) | 0/10 (0) | 1/10 (1) | 0/0 (0) | 0/0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/293 (0) | 0/292 (0) | 0/208 (0) | 0/61 (0) | 0/60 (0) | 0/42 (0) | 1/31 (1) | 0/35 (0) | 0/27 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/293 (0) | 0/292 (0) | 0/208 (0) | 0/61 (0) | 0/60 (0) | 0/42 (0) | 0/31 (0) | 1/35 (1) | 0/27 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 7 (7) | 8 (8) | 6 (7) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days